CLINICAL TRIAL: NCT03390374
Title: Oral Nystatin Prophylaxis to Prevent Systemic Fungal Infection in Very Low Birth Weight Preterm Infants: a Randomized Controlled Trial
Brief Title: Oral Nystatin Prophylaxis to Prevent Systemic Fungal Infection in Very Low Birth Weight Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Lily Rundjan, Lily Rundjan, MD, Neonatologist, Dr Cipto Mangunkusumo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 434/PT02.FK/ETIK/2010
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Fungal Infections Systemic
Keywords: Nystatin; Fungal colonization; Systemic fungal infections
MeSH Terms: interventions — Nystatin

STUDY DESIGN:
Intervention Model Description: The participants is randomly allocated into 2 study groups (nystatin group and control group) during study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nystatin group (Experimental): Nystatin oral 1 mL (0.5 mL coated in oral cavity and the rest was given through orogastric tube) three times a day
  Interventions: Drug: Nystatin Oral
- Control group (No Intervention): Sterile water 1 mL three times a day for oral hygiene

INTERVENTIONS:
Drug: Nystatin Oral — Nystatin oral suspension
  Other Names: Mycostatin
  Arms: Nystatin group

SUMMARY:
This study determines the effectiveness of oral nystatin as prophylaxis in order to prevent systemic fungal infection in very low birth weight preterm neonates. 47 participants received oral nystatin and 48 participants received sterile water as part of oral hygiene.

DETAILED DESCRIPTION:
Oral nystatin is an effective and safe alternative fungal prophylaxis. Some previous studies (1 randomized controlled trial and 4 observational studies) showed that oral nystatin prophylaxis reduce fungal colonization and decrease risk of systemic fungal infection in very low birth weight infants.

Nystatin is a non-absorbable antifungal agent with minimal side effects that works by binding on the major component of fungus cell membrane and causes death of the fungus. Its efficacy as fungal prophylaxis is comparable with Fluconazole but does not linked to drug-induced liver injury.

To determine this effectivity, we recruit eligible neonates who are admitted in our neonatal intensive care unit and randomly assign them into 2 groups once noted written parental consent. One group is given nystatin via oral and/or orogastric tube and the other group only receives sterile water as part of oral hygiene. Weekly fungal surveillance cultures (oropharyngeal and rectal) are done to evaluate colonization. Further examinations (blood/cerebrospinal fluid/deep tissue/urine culture) are done once noted clinical signs of systemic fungal infections.

Data analysis is conducted with intent-to treat approach. Significance testing is done by chi-square or fisher's exact test as needed.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <= 32 weeks and/or birth weight <=1500 grams
* 1 or more systemic fungal infection risk factors (antibiotic therapy, intravenous access, endotracheal tube, orogastric tube, urinary catheter, corticosteroid therapy, parenteral nutrition, theophylline therapy)

Exclusion Criteria:

* Suspected of having necrotizing enterocolitis within 72 hours after birth, cyanotic congenital heart disease, chromosomal defects, or critical conditions whom were not expected to live more than 72 hours after birth

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Fungal colonization | 1 to 6 weeks
  Weekly oropharyngeal and rectal fungal surveillance results are evaluated. Colonization is considered positive if yeast cells were found on either oral or rectal specimen
Systemic fungal infection | 1 to 6 weeks
  Culture of blood, cerebrospinal fluid, deep tissue, or urine is evaluated in participants with symptoms/signs of systemic infection. Proven systemic fungal infection is defined as a positive blood, cerebrospinal fluid, deep tissue, or urine culture (> 10.000 or more colony forming unit/mL from sterile bladder catheterization or suprapubic aspiration)

SECONDARY OUTCOMES:
Mortality rates | 1 to 6 weeks
  Fungal and overall related mortality rates
Nystatin-related adverse drug reactions | 1 to 6 weeks
  Any side effects of nystatin as reported in references

CONTACTS AND LOCATIONS:
Overall Officials: Lily Rundjan, MD, Principal Investigator — Dr Cipto Mangunkusumo General Hospital

REFERENCES:
- [Derived] Rundjan L, Wahyuningsih R, Oeswadi CA, Marsogi M, Purnamasari A. Oral nystatin prophylaxis to prevent systemic fungal infection in very low birth weight preterm infants: a randomized controlled trial. BMC Pediatr. 2020 Apr 17;20(1):170. doi: 10.1186/s12887-020-02074-0. PMID 32303210